CLINICAL TRIAL: NCT04781699
Title: Optimising Secondary Prevention and Quality of Life in Early Cardiac Rehabilitation
Acronym: OSPREY-CR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Hallam University (Other)
Collaborators: AstraZeneca (Industry); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Northumbria Healthcare NHS Foundation Trust (Other); NHS Ayrshire and Arran (Other); Belfast Health and Social Care Trust (Other); Aneurin Bevan University Health Board (Other)
Responsible Party: Principal Investigator, Simon Nichols, Senior Research Fellow, Sheffield Hallam University
Other Study IDs: ER22491844
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Myocardial Infarction; Acute Coronary Syndrome; Coronary Heart Disease; Heart Failure
Keywords: Cardiac Rehabilitation; Secondary Prevention; Medication Adherence; Smoking Cessation; Healthy diet; Lifestyle; Exercise; Quality of life
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Myocardial Infarction; Acute Coronary Syndrome; Coronary Disease; Heart Failure; Medication Adherence; Smoking Cessation; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this research is to explore the adherence and drop-out from early cardiac rehabilitation (CR), to inform interventions to support patient's adherence to CR and facilitate maintenance. The secondary aim is to understand which aspects of CR are essential for improving health-related quality of life in the short and long-term. This research will comprise four stages adopting a mixed-methods, quasi-experimental, repeated measures design.

DETAILED DESCRIPTION:
This study will explore the attitudes of patients and healthcare practitioners towards the components of CR (diet, smoking, and medication) and their relationship with improving patients' perceived health and wellbeing. We will apply user-centred approaches by working with patients and other stakeholders to develop the best solutions that help patients to adhere to relevant health behaviour changes. The proposed study will use a mix of surveys and interviews. This will conclude with a two-day workshop with patients and health care professionals to come up with recommendations for improving adherence to CR.

Stage 1: A bespoke survey has been designed to examine the perceptions of patients and health care professionals. The survey will include questions around, CR referral, uptake and adherence rates. Factors that hinder and improve attendance to CR will be explored. Surveys will be distributed amongst CR patients across six centres in the United Kingdom: Sheffield, London, North of England, Scotland, Wales, and Northern Ireland. The aim is to collect survey responses from 498 patients.

Stage 2: Qualitative interviews will be carried out with both patients and professionals. Topics will include factors that improve or hinder attendance and completion of CR. In addition, factors in CR which assist with improving quality of life will be explored. This will provide a more in-depth understanding of challenges to attendance identified in study 1. Up to 10 patients from each site will be interviewed, plus up to 20 health care professionals across all sites.

Stage 3: Up to 30 participants recruited across regions will be invited to take part in a two-day workshop. The two-day co-design workshop will involve patients, clinicians, CR providers, and researchers. The aim is to develop recommendations and approaches to improving attendance and completion of CR. This will include improvements to existing CR.

Study Conduct, Participant identification, inclusion, and exclusion

Each of the six sites currently delivers comprehensive early CR and provides access to patients and providers with lived experience of the core components and behaviour changes associated with CR adherence. A local principal investigator who is responsible for the leadership of a research study has been identified at each site to oversee conduct of the study protocol and facilitate participant recruitment. Participants will represent a range of demographic backgrounds including ethnicity, socioeconomic group, cardiac diagnosis and length of engagement with CR. Recruitment to interviews will stop when no new themes are being identified from the interviews (data saturation).

Healthcare professionals meeting our inclusion criteria will be approached directly, by the principal investigator at each study site. People interested in the study will be given an information sheet, and a minimum of 24 hours to consider study information before recruitment. Patients will be identified and invited to take part in the qualitative study by their healthcare professional upon referral to a CR programme.

Patients providing verbal consent will then be contacted by a member of the research team. These patients will also be invited to take part in the qualitative interviews investigating long-term adherence to CR (after six months). In the event that too few of the patients are available for the interview after six months, further patients will be retrospectively identified through the patient records kept by the CR team.

Participant consent and withdrawal

Written informed consent will be sought from participants at all stages of the study including the initial survey, subsequent interviews and/or co-design event. It will be clear at all times throughout the research that participation is voluntary and withdrawal at any stage without challenge will be supported. Information relating to participant consent will make explicit than any data collected prior to the participants' withdrawal may be retained for analysis.

Survey

Surveys will be completed online or sent via post to all identified eligible patients. If a patient decides to complete the survey online, an accessible email link will be sent via a web link using a licensed copy of Qualtrics survey software. Participants will be asked to read the study information and sign/digitally tick consent before proceeding to the survey questions.

Interviews and co-design event

Eligible participants who are interested in our study will be provided with written information sheets and offered the opportunity to ask questions by phone, email or where possible, face-to-face with the local principal investigator and/or a member of the core research team at Sheffield Hallam University. Participants will be given a minimum of 24 hours to consider the study information, after which time they will be contacted to arrange attendance.

Ethical considerations

Risks to participants are estimated to be low; although it is possible there may be some emotional effect of discussing issues and experiences related to cardiovascular disease, treatment, and its potential impact on quality of life. Participants will be made aware of the nature of the topics to be discussed during the informed consent process so that they know what to expect. Participants will be made aware that they can withdraw from the study at any time, or avoid any topics that cause discomfort. The co-design workshop will be facilitated in a way that fosters sharing, non-judgment, and equality amongst group members. It is important to manage expectations that group discussions during workshops are for research purposes, and not directly intended as patient support groups. Links and contact details will be provided for patients who express a need for further support, both verbally and via participant information sheets.

ELIGIBILITY:
Inclusion criteria patients:

* Patients who fall within the National Audit of CR (NACR) priority groups. These include Myocardial Infarction (MI), MI + Percutaneous Coronary Intervention (PCI), PCI, Coronary Artery Bypass Graft (CAGB), and Heart Failure.
* Aged over 18 years (i.e., all adults).
* No evidence of cognitive impairment which will limit the ability to follow basic instructions.

Inclusion criteria professionals:

* Those who have a key responsibility for delivering or managing CR at one of the six local sites, including - healthcare professionals and/or CR providers.

Exclusion criteria patients:

* Patients who fall outside of the NACR priority groups.
* Aged under 18 years (i.e., all adults).
* Evidence of cognitive impairment which will limit the ability to follow basic instructions (Participants unable to give informed consent).

Exclusion criteria professionals:

* Trainee or administrative staff members.
* Staff members with less than four months of experience working in CR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include patients and health care professionals across six CR sites across the UK who currently delivers comprehensive early CR. Each site will provide access to patients and providers with lived experience of the core components and behaviour changes associated with CR adherence. A local Principal Investigator has been identified at each site to oversee the local conduct of the study protocol and facilitate participant recruitment. A purposive sampling approach for the qualitative interveiws will be employed to ensure that participants represent a range of demographic backgrounds including ethnicity, socioeconomic group, cardiac diagnosis and length of engagement with CR.
Sampling Method: Probability Sample
Enrollment: 498 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Reasons people attend early cardiac rehabilitation (quantitative method). | Start of cardiac rehabilitation
  Using a pre-developed questionnaire.
Attendance to early cardiac rehabilitation | End of cardiac rehabilitation ~ 8 weeks.
  Measured by number of patients referred to cardiac rehabilitation and proportion who take up cardiac rehabilitation.
Reasons people adhere to early cardiac rehabilitation (quantitative method). | End of cardiac rehabilitation ~ 8 weeks
  Using a pre-developed questionnaire.
Reasons people adhere to cardiac rehabilitation (qualitative method). | End of cardiac rehabilitation ~ 8 weeks
  Using a semi-structured qualitative interview.
Reasons people adhere to core components of cardiac rehabilitation (quantitative method). | 6 months after completion of cardiac rehabilitation
  Using a pre-developed questionnaire.
Reasons people adhere to components of cardiac rehabilitation in the long term (qualitative method). | 6 months after completion of cardiac rehabilitation
  Using a semi-structured qualitative interview.
Reasons people drop-out of cardiac rehabilitation (quantitative method). | End of cardiac rehabilitation ~ 8 weeks
  Using a pre-developed questionnaire.
Reasons people drop-out of cardiac rehabilitation (quantitative method). | 6 months after completion of cardiac rehabilitation
  Using a pre-developed questionnaire.
Drop-out of early cardiac rehabilitation (quantitative method) | End of cardiac rehabilitation ~ 8 weeks.
  Drop-out will be defined as attending less than 50% of sessions.
Reasons people drop-out of early cardiac rehabilitation (qualitative method) | End of cardiac rehabilitation ~ 8 weeks.
  Using a semi-structured qualitative interview.

SECONDARY OUTCOMES:
Patient perceptions on which components of cardiac rehabilitation improve health related quality of life (quantitative method). | Start of cardiac rehabilitation
  Using a pre-developed questionnaire.
Patient perceptions on which components of cardiac rehabilitation improve health related quality of life (quantitative method). | End of cardiac rehabilitation ~ 8 weeks
  Using a pre-developed questionnaire.
Patient perceptions on which components of cardiac rehabilitation improve health related quality of life (quantitative method). | 6 months after completion of cardiac rehabilitation
  Using a pre-developed questionnaire.
Patient perceptions on which components of cardiac rehabilitation improve health related quality of life (qualitative method). | End of cardiac rehabilitation ~ 8 weeks
  Using a semi-structured qualitative interview.
Patient perceptions on which components of cardiac rehabilitation improve health related quality of life (qualitative method). | 6 months after completion of cardiac rehabilitation
  Using a semi-structured qualitative interview.
Professional perspectives of supporting adherence to core components of cardiac rehabilitation (qualitative method). | Within 5 months from study start date.
  Using a semi-structured qualitative interview.

OTHER OUTCOMES:
Intervention development | 10 months after study start date
  Via a co-design event with patients and healthcare professionals to create a clear description of an intervention package. This is based on factors reported from the primary and secondary outcome measures.

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne, Blyth
  - Aneurin Bevan University Health Board, Ystrad Mynach, Gwent
  - Royal Brompton Hospital, London, Harefield Middlesex
  - Sheffield Teaching Hospitals, Sheffield, South Yorkshire
  - Belfast Health and Social Care Trust, Belfast
  - NHS Ayrshire and Arran, Kilmarnock

IPD SHARING:
Plan to Share IPD: Undecided